CLINICAL TRIAL: NCT01493882
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Multicenter, Parallel Group, 2-Part Study of JNJ-39758979 in Symptomatic Adult Subjects With Uncontrolled, Persistent Asthma
Brief Title: Study of JNJ-39758979 in Symptomatic Adult Patients With Uncontrolled Asthma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was withdrawn due to 2 cases of agranulocytosis in a different clinical trial with this same drug.
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: DIRECTOR CLINICAL DEVELOPMENT, Janssen R&D US
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR100710; 39758979ASH2002 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.); 2011-003852-37 (EudraCT Number)
Record Dates: First submitted 2011-12-15; First posted 2011-12-16 (Estimated); Last update posted 2012-05-14 (Estimated); Status verified 2012-05

CONDITIONS: Asthma
Keywords: Uncontrolled Persistent Asthma, Dyspnea, Wheezing
MeSH Terms: conditions — Asthma; Dyspnea; Respiratory Sounds

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- JNJ-39758979 30 mg/d (Experimental)
  Interventions: Drug: JNJ-39758979 30 mg/d
- JNJ-39758979 100 mg/d (Experimental)
  Interventions: Drug: JNJ-39758979 100 mg/d
- JNJ-39758979 300 mg/d (Experimental)
  Interventions: Drug: JNJ-39758979 300 mg/d

INTERVENTIONS:
Drug: Placebo — Form = tablet, route = oral administration, once daily from Week 0 to Week 24 for Part 1 and Part 2
  Arms: Placebo
Drug: JNJ-39758979 30 mg/d — Unit = mg, number = 30, form = tablet, route = oral administration, once daily from Week 0 to Week 24 only for Part 2
  Arms: JNJ-39758979 30 mg/d
Drug: JNJ-39758979 100 mg/d — Unit = mg, number = 100, form = tablet, route = oral administration, once daily from Week 0 to Week 24 only for Part 2
  Arms: JNJ-39758979 100 mg/d
Drug: JNJ-39758979 300 mg/d — Unit = mg, number = 300, form = tablet, route = oral administration, once daily from Week 0 to Week 24 for Part 1 and Part 2
  Arms: JNJ-39758979 300 mg/d

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and tolerability of JNJ-39758979 compared with placebo in patients with uncontrolled asthma despite current treatment with inhaled corticosteroids and/or long-acting beta 2-agonist (LABA) and/or montelukast for at least 4 weeks.

DETAILED DESCRIPTION:
This is a two-part study; each part of the study (Part 1 and Part 2) will be approximately 34 weeks in duration including a 4-week screening phase, a 24-week placebo-controlled treatment phase and a six-week follow-up phase. In Part 1, patients will be randomly assigned to receive placebo or JNJ-39758979 300 mg once daily through Week 24. In Part 2, patients will be randomly assigned to 1 of 4 treatment groups to receive treatment with placebo, 30 mg, 100 mg, or 300 mg of JNJ-39758979 once daily through Week 24. Safety assessments and evaluations to determine the efficacy of JNJ-39758979 to reduce the signs and symptoms of asthma will be performed both on a daily basis via electronic diary and at study visits.

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of asthma for at least 6 months before screening. -Has been receiving inhaled corticosteroids (≤ 1000 µg fluticasone or its equivalent) alone or in conjunction with long-acting Beta 2-agonist (salmeterol, formoterol, etc.) and/or montelukast.
* Have an ACQ score ≥ 1.5 at screening. - Must be healthy and medically stable on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening
* Must be post-menopausal or if pre-menopausal, must use an acceptable method of birth control.

Exclusion Criteria:

* Has ever had a life-threatening asthma attack including respiratory arrest, intubation, or intensive care unit admission due to asthma. -Has a history of any other chronic respiratory condition including chronic obstructive pulmonary disease, bronchiolitis, bronchiectasis, allergic bronchopulmonary aspergillosis (mycosis), occupational asthma, sleep apnea or pulmonary hypertension.-Has initiated or discontinued allergen immunotherapy within 12 weeks of screening. -Has smoked within 3 years of screening or has a history of smoking ≥ 10 pack years (1 pack year = 20 cigarettes smoked per day for 1 year) or equivalent, or a positive urine cotinine test at Screening. -Has any known malignancy or has a history of malignancy with the exceptions of basal cell carcinoma or squamous cell carcinoma. -Has chronic or recurrent infectious disease, including, but not limited to: active tuberculosis.-Has a clinically significant, acute respiratory infection within 4 weeks of screening. -Has had a substance abuse (drug or alcohol) problem within the previous 3 years.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-03; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
The absolute change from baseline in percent-predicted prebronchodilator forced expiratory volume (FEV1) at Week 16 in Part 1 and in Part 2. | Baseline, Week 16

SECONDARY OUTCOMES:
Change from baseline in Asthma Control Questionnaire (ACQ) at Week 16 in Part 1 and Part 2 | Baseline, Week 16
Change from baseline in postbronchodilator percent-predicted forced expiratory volume in 1 second (FEV1) at Week 16 in Part 1 and Part 2 | Baseline, Week 16
Change from baseline in daytime asthma diary symptom score at Week 16 in Part 1 and Part 2 | Baseline, Week 16
Change from baseline in nighttime asthma diary symptom score at Week 16 in Part 1 and Part 2 | Baseline, Week 16
Change from baseline in average rescue medication use at Week 16 in Part 1 and Part 2 | Baseline, Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.